CLINICAL TRIAL: NCT02355236
Title: A Prospective, Randomized, Double-blinded, Double-dummy, Active-controlled, Multi-center, Interventional Study to Compare Gastro-protective Effect and Pain Relief Effect of Naxozol Compared to Celecoxib in Patients With Osteoarthritis
Brief Title: Gastro-protective Effect and Pain Relief Effect of Naxozol Compared to Celecoxib in Patients With Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Seong-Hwan Moon, Professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Naxozol_P4_1
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: Naxozol; LDQ; GSRS; Osteoarthritis; Gastroprotective
MeSH Terms: conditions — Osteoarthritis | interventions — Naproxen; Omeprazole; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental): Naproxen/Esomeprazol 500/20mg and Comparator-Placebo for 12 weeks
  Interventions: Drug: Naproxen/Esomeprazol 500/20mg; Drug: Comparator-Placebo
- Comparator Group (Active Comparator): Celecoxib 200mg and Naxozol-Placebo for 12 weeks
  Interventions: Drug: Celecoxib 200mg; Drug: Naxozol-Placebo

INTERVENTIONS:
Drug: Naproxen/Esomeprazol 500/20mg — Tablet, b.i.d.
  Other Names: Naxozol
  Arms: Test Group
Drug: Celecoxib 200mg — Capsule, o.d.
  Other Names: Celebrex
  Arms: Comparator Group
Drug: Naxozol-Placebo — Tablet (which is identical to Naxozol), b.i.d.
  Arms: Comparator Group
Drug: Comparator-Placebo — Capsule (which is identical to Celebrex), o.d.
  Arms: Test Group

SUMMARY:
Naxozol is a combination product of naproxen, a non-steroidal anti-inflammatory drug (NSAID) and esomeprazole, a proton pump inhibitor which is designed to improve symptoms and reduce risk of gastric ulcers in patients at risk of developing NSAID-associated gastric ulcers in the treatment of osteoarthritis, rheumatoid arthritis, and ankylosing spondylitis. The purpose of this study is to investigate whether naxozol protects the gastrointestinal tract effectively compared to celecoxib, a COX-2 inhibitor.

DETAILED DESCRIPTION:
A total of 10 orthopedic investigators will participate in this study. The effectiveness in gastro-protection of study drug will be assessed by Leeds Dyspepsia Questionnaire (LDQ). The orthopedic investigators will be trained with this questionnaire administration by an expert gastroenterologist prior to starting this study.

ELIGIBILITY:
Inclusion Criteria:

* Koreans given informed consent
* Patients who have ability of reading comprehension and completing questionnaires (EQ-5D and VAS)and have willingness to follow-up 12 weeks
* Patients with osteoarthritis symptoms confirmed by his/her medical history and with pain-VAS of 40 and more

Exclusion Criteria:

* Patients who participate into other interventional study or had participated within 30 days before screening
* Alcohol or drug abuse within 6 months or alcohol consumption of 21 units and more in a week
* Peptic ulcers accompanied with a complication such as bleeding, perforation, penetration or gastric outlet obstruction within 5 years, or a history of active peptic ulcer or peptic ulcer without a complication within 6 months at screening
* Patients who are known with Helicobacter pylori infection but have not received any bacteriostatic treatment
* Known gastroesophageal reflux disease (GERD)
* Any following joint diseases which may significant effect to the efficacy and safety assessments: septic arthritis, inflammatory joint arthritis such as rheumatoid arthritis, gout, recurrent pseudo-pain, Paget's disease, joint fracture, joint ochronosis, acromegaly, hematochromatosis, Wilson's disease, primary osteochondrosis, Ehlers Danlos Syndrome, or other collagen genetic disorder
* Patients who are scheduled admissions to hospital for elective surgery during this study
* History of gastrointestinal cancer
* Gastrointestinal disorders related to drug malabsorption
* Gastrointestinal bleeding, cerebral bleeding, other bleeding disorders, or severe hematological disorders
* Clinically significant diseases such as moderate or severe liver diseases (Child Pough Class II or more), severe heart failure or a history of coronary artery bypass graft (CABG), severe kidney diseases (CrCl<30ml/min)
* Know allergy experiences with any ingredient of study drugs or with other NASIDs or protocol pump inhibitors (PPIs)
* Patients who had had a joint surgery for osteoarthritis within 1 year
* Women of childbearing potential who do not agree with clinically appropriate contraception during this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Leads Dyspepsia Questionnaire (LDQ) Change | Baseline, 12 weeks
  Mean change from baseline of Leads Dyspepsia Questionnaire

SECONDARY OUTCOMES:
Mean LDQ | Baseline, 12 weeks
  Mean value of Leads Dyspepsia Questionnaire at 12 weeks
Gastrointestinal Symptom Rating Scale (GSRS) Change | Baseline, 12 weeks
  Mean change from baseline of Gastrointestinal Symptom Rating Scale
Gastrointestinal Adverse Events Rate | Baseline, 12 weeks
  Dyspepsia, Diarrhoea, Nausea, Abdominal Pain, Heartburn
Drug Discontinuation Rate Due to Gastrointestinal Adverse Events | Baseline, 12 weeks
Pain Relief Effect, mean change from baseline of Pain Visual Analogue Scale (VAS) | Baseline, 12 weeks
  Mean change from baseline of Pain Visual Analogue Scale (VAS)
Quality of Life Change, mean change from baseline of EQ-5D | Baseline, 12 weeks
  Mean change from baseline of EQ-5D
Treatment Compliance | Baseline, 12 weeks
  Non-compliance is defined less than 80%
Rescue Drugs Usage | Baseline, 12 weeks
  Acetaminophen ER 650mg and/or Almagate 500mg will be administrated for control of severe pain events and/or of severe gastrointestinal events.
Adverse Events | Baseline, 12 weeks
  Adverse Events and Abnormalities from Vital Signs, Physical Exam, and Clinical Laboratories

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hwan Moon, M.D., Ph.D., Study Chair — Severance Hospital
Locations (10):
- South Korea (10):
  - Hallym University Medical Center, Anyang-si
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul